CLINICAL TRIAL: NCT07358884
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of QLS5316 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: First in Human Study of QLS5316 in Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS5316-101
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors; Colorectal Cancer; Gastric Cancer or Gastroesophageal Junction Adenocarcinoma; Head and Neck Squamous Cell Carcinoma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS5316 (Experimental): patients with advanced solid tumors were administrated with varying doses of QLS5316 specified in protocol
  Interventions: Drug: QLS5316

INTERVENTIONS:
Drug: QLS5316 — Varying doses of QLS5316

SUMMARY:
This is a first-in-human (FIH) Phase I, multi-center, open-label, study of QLS5316, in patients with advanced solid tumors. The study aim to evaluating the safety, tolerability, preliminary efficacy, pharmacokinetics (PK), and immunogenicity of QLS5316 as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1
3. Life expectancy ≥ 3 months;
4. Measurable disease per RECIST v1.1
5. Adequate organ and marrow function as defined in the protocol
6. Dose escalation and PK expansion stages: Histologically or cytologically confirmed locally advanced or metastatic malignant solid tumors that cannot undergo radical surgery or radiotherapy, who have failed SOC or SOC is not available
7. Cohort expansion stage: Patients with histologically or cytologically confirmed locally advanced or metastatic malignant solid tumors that cannot undergo radical surgery or radiotherapy, including CRC, GC/GEJ, HNSCC (mouth, oropharynx, hypopharynx or larynx), EGFR-sensitive mutant NSCLC and EGFR wild-type NSCLC or other advanced malignant solid tumors who have failed SOC or SOC is not available.

Exclusion Criteria:

1. Prior treatment with antibody-drug conjugates (ADCs) containing topoisomerase I inhibitors, or prior treatment with EGFR and/or c-MET targeted ADCs
2. Untreated or active brain metastasis
3. Presence of Grade ≥ 2 toxicity (according to the Common Terminology Criteria for Adverse Events (CTCAE Version 5.0) ) left over from prior therapy
4. Patients with a history of interstitial lung disease (ILD)/non-infectious pneumonia, or patients whose suspected ILD/non-infectious pneumonia cannot be ruled out by imaging examination at screening; patients with radiation pneumonitis who do not require steroid treatment are allowed to be enrolled;
5. Patients with a history of active tuberculosis, active autoimmune diseases or autoimmune diseases that may recur
6. Patients with a history of severe cardiovascular and cardiovascular diseases
7. Clinically uncontrollable third space effusion
8. Presence of persistent uncontrolled systemic bacterial, fungal or viral infections or severe infections within 4 weeks before the first dose in the study, or active infections requiring systematic antibiotic treatment within 1 week before the first dose in the study;
9. Known hypersensitivity reactions or delayed-type sensitization to some components or analogues of the investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by NCI-CTCAE v5.0 | From time of Informed Consent to 30 days post last dose of QLS5316
  To evaluate the safety and tolerability of QLS5316
Number of Participants With Clinical Laboratory Test Abnormalities | From time of Informed Consent to 30 days post last dose of QLS5316
  Clinical laboratory test included Hematology, Blood and serum chemistry, Coagulation function, and Fecal occult blood.
12-lead ECG(Including heart rate, QT interval, QTc interval, and P-R interval) | From time of Informed Consent to 30 days post last dose of QLS5316
  Assessment of abnormal electrocardiogram parameters before and after treatment
Number of participants with physical examination abnormalities | From time of Informed Consent to 30 days post last dose of QLS5316
  Including general conditions, skin and mucosa, systemic superficial lymph nodes, head and neck, chest, abdomen, spine and extremities, nervous system, and other examinations.
Number of participants with vital signs abnormalities | From time of Informed Consent to 30 days post last dose of QLS5316
  Including body temperature, respiratory rate, pulse, blood pressure, and oxygen saturation
DLT | From time of first dose of QLS5316 to end of DLT period (21 days)
  Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Protocol
MTD | 1 year
  the maximum tolerated dose (MTD) or maximum administered dose (MAD, if MTD fails to be determined) of QLS5316 monotherapy
RP2D | 2 year
  the recommended phase II dose of QLS5316 monotherapy